CLINICAL TRIAL: NCT02886650
Title: Impact of Thermocoagulation During Invasive EEG Monitoring in Children With Focal Drug-resistant Epilepsies
Acronym: COAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCX_2015_31
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
Keywords: Paediatrics; epilepsy surgery; genetic mutation; focal seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Electrocoagulation

ARMS (1):
- Thermocoagulation (Experimental)
  Interventions: Procedure: Thermocoagulation

INTERVENTIONS:
Procedure: Thermocoagulation — Thermocoagulation During pre-surgical Invasive EEG Monitoring

SUMMARY:
When focal epilepsies become drug-resistant, it could be eligible for cortical surgical resection. Therefore, an invasive EEG monitoring with depth electrodes is often needed during presurgical evaluation. Some of these children can have access to thermocoagulation inside the ictal onset zone, at the end of the monitoring and before to remove the electrodes. These thermocoagulations can disorganize the epileptogenic network thanks to millimetric cortical lesions around the electrodes. The aim is to stop or at least, to reduce the seizure frequency for few weeks or months. This could be a benefit for the child, and also a confirmation of the ictal onset zone and guide the surgeon. This technique is currently used in adult population for years, but remains very rare in children.

ELIGIBILITY:
Inclusion Criteria:

* age 18 month to 17 years old
* focal drug-resistant epilepsy
* small size lesion (1 or 2 gyri) or cryptogenic epilepsy
* indication for EEG monitoring with depth electrodes during presurgical evaluation

Exclusion Criteria:

* formal contraindication to surgery or anaesthesia
* functional area or potentially large epileptic area
* refusal to participate in the study
* no health insurance coverage

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Number of children with a decrease of at least 50% of the seizure frequency | one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde CHIPAUX, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France